CLINICAL TRIAL: NCT02396810
Title: A Single-center, Prospective, Randomized Controlled Trial Investigating the Utility if Intraoperative MRI in Transphenoidal Pituitary Surgery Off Macroadenomas.
Brief Title: Utilization of iMRI for Transsphenoidal Resection of Pituitary Macroadenomas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending additional funding
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Nathan E. Simmons, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUDY00028376 D14236
Record Dates: First submitted 2015-03-05; First posted 2015-03-24 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Pituitary Macroadenoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intra-operative MRI (Placebo Comparator): Patients undergo transsphenoidal surgery without an intra-operative MRI.
  Interventions: Procedure: Transsphenoidal resection of pituitary macroadenoma
- intra-operative MRI (Experimental): Patients undergo transspheonidal surgery followed by intra-operative MRI.
  Interventions: Other: intra-operative MRI; Procedure: Transsphenoidal resection of pituitary macroadenoma

INTERVENTIONS:
Other: intra-operative MRI — Intra-operative magnetic resonance imaging under general anesthesia
  Arms: intra-operative MRI
Procedure: Transsphenoidal resection of pituitary macroadenoma — Routine transsphenoidal resection of pituitary macro adenomas

SUMMARY:
The investigators are studying the utility of intra-operative magnetic resonance imaging (iMRI) during transsphenoidal pituitary surgery for large macroadenomas by randomizing patients to either an intra-operative MRI after resection, or no intra-operative MRI. The investigators will then count the number of gross total resection in each group of patients and also the complications related to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-90
* Capable of giving informed consent
* Elect for transsphenoidal surgery
* Has pre-operative MRI demonstrating pituitary tumor that is:

  1. deemed resectable using a transsphenoidal approach and
  2. has a maximal diameter equal to or greater than 15 mm.
* No contraindications for MRI.

Exclusion Criteria:

* Children (age < 18)
* Not able to give consent
* No pituitary tumor visible on MRI or an adenoma measuring less than 15mm in maximal dimension.
* Unable to tolerate MRI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of gross total or maximal resection | 24 hours after surgery
  Determine whether use of iMRI in transsphenoidal pituitary surgery for pituitary macroadenomas significantly increases the rate of maximal resection

SECONDARY OUTCOMES:
Operative time | intraoperative
  Length of operation
Frequency of post-operative CSF leak | 30 days post surgery
  Frequency of post-operative Cerebrospinal Fluid (CSF) leak
Rate of Readmission | 30 days post surgery
  Frequency of readmission
Length of anesthesia time | intraoperative
  Length of time participant is under anesthesia
Rate of post-operative endocrinopathies | 30 days post surgery
  Rate of post-operative endocrinopathies

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States